CLINICAL TRIAL: NCT00924859
Title: The Role of Factor XIII Activation Peptide and D-dimer Values for the Diagnosis of Cerebral Venous Thrombosis
Brief Title: The Role of Factor XIII Activation Peptide and D-dimer Values for the Diagnosis of Cerebral Venous Thrombosis (CVT)
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Schweizerische Herzstiftung (Other)
Responsible Party: Departement of Neurology, Inselspital Bern, Universitiy Hospital
Other Study IDs: 112/09
Record Dates: First submitted 2009-06-15; First posted 2009-06-19 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Cerebral Venous Thrombosis
Keywords: cerebral venous thrombosis; stroke; coagulation
MeSH Terms: conditions — Intracranial Thrombosis; Stroke; Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with clinical suspicion of CVT
  Interventions: Other: ELISA Test

INTERVENTIONS:
Other: ELISA Test — assess the overall accuracy of D-dimer values and FXIII activation peptide (FXIII-AP), using a newly developed ELISA test

SUMMARY:
The investigators aim to assess the overall accuracy of D-dimer values and FXIII activation peptide (FXIII-AP), using a newly developed ELISA test, to exclude CVT in patients with clinical suspicion of CVT.

DETAILED DESCRIPTION:
Background

Because of the broad clinical spectrum it is often difficult to establish the diagnosis of cerebral venous thrombosis (CVT). Combined MRI/MRV and contrast-enhanced CT are the most accurate methods for diagnosis of CVT. However these methods are often not available on an emergency basis. This stresses the need for additional widely available tests such as coagulation markers to exclude CVT. The diagnostic value of D-dimer levels for the exclusion of CVT is still under debate. Other potential coagulation markers have not been systematically investigated. The investigators aim to assess the overall accuracy of D-dimer values and FXIII activation peptide (FXIII-AP), using a newly developed ELISA test, to exclude CVT in patients with clinical suspicion of CVT. Consecutive patients with clinical suspicion of CVT at the emergency department of the University Hospital Bern will be included in this study over a two year period. All included patients will receive standard care applied by the treating physician who will follow international recommendations. Patient involvement in the study shall not influence any treatment decision. On admission patients will undergo a complete diagnostic work-up, including a clinical neurological examination, standard laboratory examination including D-dimer values, and brain contrast CT and/or MRI/MRV. In addition, plasma FXIII-AP will be analyzed. FXIII-AP will be analyzed at the Hemostasis Research Laboratory, Department of Hematology, University of Bern, based on a newly developed highly sensitive and specific ELISA method. The investigators will be blinded for the clinical symptoms and diagnosis of the patient. The study will be conducted according to the guidelines of the STARD (Standards for Reporting Diagnostic Accuracy) initiative.

The following primary evaluation criteria will be analysed:1) The overall diagnostic accuracy of FXIII-AP to exclude CVT in patients with clinical suspicion of CVT; 2) The overall diagnostic accuracy of D-dimer to exclude CVT in patients with clinical suspicion of CVT; 3) Roc curves will be calculated.

Prespecified subgroup analyses will be performed according to the clinical presentation: 1) isolated headache; 2) isolated intracranial hypertension (headache and papilledema); 3) Focal neurological deficits and/or seizures and/or disturbances of consciousness. Furthermore, prespecified subgroup analyses will be performed according to modes of onset: 1) acute (symptoms < 48 hours duration); 2) subacute (symptoms > 48 hours and < 7 days duration); 3) chronic (symptoms > 7 days duration).

The following secondary evaluation criteria will be assessed: 1) The overall frequency of CVT in patients with clinical suspicion of CVT; 2) The overall frequency of other diseases in patients with clinical suspicion of CVT; 3) The site of involved veins and sinus in patients with CVT.

Objective

The investigators aim to assess the overall accuracy of D-dimer values and FXIII activation peptide (FXIII-AP), using a newly developed ELISA test, to exclude CVT in patients with clinical suspicion of CVT.

Methods

Consecutive patients with clinical suspicion of CVT at the emergency department of the University Hospital Bern will be included in this study over a two year period. All included patients will receive standard care applied by the treating physician who will follow international recommendations. D-dimer measurement at entry will be performed using a rapid sensitive assay. FXIII-AP will be analyzed at the Hemostasis Research Laboratory, Department of Hematology, University of Bern based on a highly sensitive and specific ELISA method.The investigators will be blinded for the clinical symptoms and diagnosis of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Adults with clinical suspicion of CVT
* Isolated unexplained headache of less than 30 days duration
* Headache associated with focal central neurological deficits of less than 30 days duration
* Headache associated with disturbed consciousness of less than 30 days duration
* Headache associated with epileptic seizures of less than 30 days duration
* Unexplained papilledema of less than 30 days duration

Exclusion Criteria

* Deep venous thrombosis within 3 months prior to admission
* Pulmonary embolism within 3 months prior to admission
* Ischemic stroke within 3 months prior to admission
* Myocardial infarction within 3 months prior to admission
* Other vascular disease within 3 months prior to admission
* Headache due to trauma
* Malignant neoplasia
* Treatment with anticoagulants prior to admission

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with clinical suspicion of CVT at the emergency department of the University Hospital (tertiary care clinic)
Sampling Method: Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
The overall diagnostic accuracy of FXIII-AP an D-dimer to exclude CVT in patients with clinical suspicion of CVT | at hospital entry

SECONDARY OUTCOMES:
The overall frequency of CVT in patients with clinical suspicion of CVT | at hospital entry
The overall frequency of other diseases in patients with clinical suspicion of CVT | at hospital entry
The site of involved veins and sinus in patients with CVT | at hospital entry

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Arnold, MD Prof., Principal Investigator — Dep. of Neurology, Bern University Hospital
Locations (2):
- Department of Neurology, Academic Medical Centre, University of Amsterdam, Amsterdam, Netherlands
- Dep. of Neurology, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Derived] Heldner MR, Zuurbier SM, Li B, Von Martial R, Meijers JCM, Zimmermann R, Volbers B, Jung S, El-Koussy M, Fischer U, Kohler HP, Schroeder V, Coutinho JM, Arnold M. Prediction of cerebral venous thrombosis with a new clinical score and D-dimer levels. Neurology. 2020 Aug 18;95(7):e898-e909. doi: 10.1212/WNL.0000000000009998. Epub 2020 Jun 23. PMID 32576633